CLINICAL TRIAL: NCT04674384
Title: A Randomised Feasibility Trial of an Intermittent Low Energy Diet (ILED) and Continuous Low Energy Diet (CLED) in Patients With Type 1 Diabetes and Obesity
Brief Title: Manchester Intermittent and Daily Diet Type 1 Diabetes App Study (MIDDAS-Type 1)
Acronym: MIDDAS T1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B01030
Record Dates: First submitted 2020-12-09; First posted 2020-12-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Type 1 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Low Energy Diet (ILED) (Active Comparator)
  Interventions: Dietary Supplement: Optifast meal replacement shakes
- Continuous Low Energy Diet (CLED) (Active Comparator)
  Interventions: Dietary Supplement: Optifast meal replacement shakes

INTERVENTIONS:
Dietary Supplement: Optifast meal replacement shakes — Optifast® is provided as 53g sachet. Each sachet replaces one meal. It is available in 5 flavours: vanilla, strawberry, chocolate and coffee shakes and vegetable soup.

SUMMARY:
To assess the safety, acceptability and feasibility of testing Intermittent Low Energy Diet (ILED) and Continuous Low Energy Diet (CLED) programmes for 12 weeks in a real life setting with people with T1D and obesity.

DETAILED DESCRIPTION:
The study described herein is a small randomised, open-label, single centre feasibility study of 12 patients with T1D and obesity. The aim of the study is to assess the safety, acceptability and feasibility of ILED (850kcal/day 2 days/week) and CLED (850kcal/day) over 12 weeks in a real life setting with people with T1D and obesity to help them lose weight and improve their glycaemic control. The low energy diets will involve Nestle Optifast® meal replacements as a total diet replacement (TDR).

People with T1D are becoming increasingly accustomed to remote monitoring of their blood glucose by health professionals using several continuous glucose monitoring devices including the Freestyle Libre® flash glucose monitoring system. The Freestyle Libre® allows healthcare professionals to view patient blood glucose trends and patterns from the web-based platform Libreview®. The study described herein will also assess the safety and practicality of providing remote follow-up support by healthcare professionals (dietitian, nurse and psychologist) to patients with T1D and obesity during the course of implementing the low energy diets. High-frequency remote follow up has been shown to be superior to low-frequency face-to-face care in weight management interventions. Remote care reduces participants' burden to attend face-to-face appointments and may be cost-effective compared with face-to-face care whilst improving access to care. The study described herein will incorporate high-frequency remote follow up via telephone and/or the Oviva® smartphone application facilitating messaging, video calls and self-monitoring of weight and blood pressure. The Freestyle Libre® flash glucose monitoring system will facilitate remote review of blood glucose readings.

Positive results from this feasibility study of two different low energy diets will inform whether one or both diets go forward into a large and longer term randomised efficacy trial following the Medical Research Council complex intervention guidance. This could provide the evidence base to inform the use of low energy diets in individuals with T1D and obesity for weight loss to improve their metabolic status and reduce the risk of cardiovascular and other physical and mental co morbidities associated with T1D.

ELIGIBILITY:
Inclusion Criteria:

* T1D for 12 months or longer
* HbA1c 53-108 mmol/mol
* BMI ≥ 30 kg/m2 and <50kg/ m2 or ≥27.5 kg/ m2 and <50kg/ m2 in high-risk minority ethnic groups i.e. South Asian, Black African and African Caribbean
* Multiple daily injections (MDI) or continuous subcutaneous insulin infusion (CSII)
* Completed Dose Adjustment For Normal Eating (DAFNE) education
* Access to a Freestyle Libre handset and sensors to monitor blood glucose
* Willing to use the Freestyle Libre® flash glucose monitoring system to monitor blood glucose (flash and capillary) and blood ketones and to record carbohydrate and insulin.
* Access to and ability to use a telephone. If no access to a smartphone running iOS or Android (to view the LibreLink app®) then access to a computer (to upload results to the LibreView website).
* Willing to undertake Optifast® LEDs and have previously sampled Optifast®.
* Negative urine pregnancy test at screening and agreement to maintain contraception or abstinence for the trial (where appropriate)
* Ability to read, understand and communicate in English.

Exclusion Criteria:

* Evidence of severe hypoglycaemia in the last 12 months (more than one episode requiring third party assistance) or hypoglycaemia unawareness.
* Patients with non-stable retinopathy, or grade R2 or later, or had no retinopathy screen within 12 months.
* Patients who lack capacity or are unable to read or understand written or verbal instructions in English or those diagnosed with learning difficulties.
* Confirmed pregnant via a pregnancy test at screening, planning pregnancy in the next 3 months, or currently breast feeding.
* Participants who are currently on treatment with Orlistat or other pharmacological treatments for weight loss e.g. Glucagon-like-peptide-1 (GLP-1).
* Participants who are currently taking a Sodium-Glucose Co-Transporter-2 (SGLT2) inhibitor.
* Diagnosed Gastroparesis.
* Participants who have previously had bariatric surgery for weight loss including gastric bypass and sleeve gastrectomy.
* Patients who are on chronic use of steroids (more than 20mg daily of prednisolone or its equivalent).
* Patients with known hypersensitivity to any of the ingredients of Optifast® e.g. fish, milk, soy.
* Taking prohibited medications (see Appendix 3) including warfarin or novel anticoagulants (NOAC), low molecular weight heparin (LMWH) or equivalent anti-coagulants and anti-psychotic medication or other psychotropic medications that may cause excessive weight gain.
* Substance abuse or harmful alcohol use as indicated by a score of 16 or above on the Alcohol Use Disorders Identification Test (AUDIT).[36]
* Participants with a diagnosed eating disorder, or patients with severe binge eating assessed by a score of 27 or more on the Binge Eating Scale (BES).[37]
* Participants with severe depression assessed by a score of 15 or more on the Patient Health Questionnaire-9 (PHQ-9) questionnaire.[29]
* Participants with severe anxiety assessed by a score of 15 or more on the General Anxiety Disorder (GAD-7) questionnaire.[28]
* Participants with very low self-efficacy assessed by a score of 35 or less on the Weight Efficacy Lifestyle Questionnaire (WEL-SF).[30]
* Participants with severe loss of renal function (eGFR < 30mL/min/1.73m2).
* Participants with psychiatric or physical comorbidity or scheduled for major surgery, which in the opinion of the treating medical physician, Chief Investigator (CI) or Multidisciplinary Team (MDT) would compromise their safety or adherence to the study.
* Unsatisfactory use of the Freestyle Libre® flash glucose monitoring system or unsafe use of DAFNE/insulin adjustment principles during the 14-day "run-in" period that in the opinion of the medical team may undermine the participant's safety on the trial. This includes flash and capillary monitoring of blood glucose and ketone testing.
* Patients who are currently participating in a diabetes drug trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of episodes of severe hypoglycaemia i.e. capillary blood glucose < 3.0 mmol/l or requiring 3rd party assistance or any episodes of nocturnal hypoglycaemia <3.0 mmol/l. | 14 week duration of study
Time spent in target (3.9-10mmol/l), below target (<3.9mmol/l and <3.0mmol/l) and above target (>10 mmol/l) on the Freestyle Libre® flash glucose monitoring system over 12 weeks. | 14 week duration of study
Number of episodes of Diabetic Ketoacidosis (DKA) and blood ketone β-hydroxybutyrate levels above 1.0mmol/l. | 14 week duration of study
Occurrence of Serious Adverse Events (SAEs) deemed potentially related to the dietary programmes. | 14 week duration of study

SECONDARY OUTCOMES:
Uptake to the trial i.e. percentage of those invited who are eligible and interested to take part | 14 week duration of study
Number of participants who complete the trial measured by attendance at the 12 week appointment (for ILED and CLED) | 14 week duration of study
Adherence to blood glucose and ketone monitoring i.e. frequency of capillary blood tests and scans | 14 week duration of study
Percentage of low energy days completed (for ILED and CLED) | 14 week duration of study
Dietary intake (7 day food diary). Food diaries will be analysed using Nutritics nutrition analysis software to estimate energy, fat, saturated fat, carbohydrate and protein intake | 14 week duration of study
Anonymous patient evaluation of the dietary programmes using an end of study questionnaire | 14 week duration of study
  The End of Study Questionnaire will be analysed using appropriate descriptive statistics for closed questions (scales 1 to 10 with 1 indicating "not at all" and 10 indicating "extremely" in the context of questions around satisfaction, ease of completion etc.). Key themes will be extracted without formal analysis from open questions to inform future research.
Percentage of multi-disciplinary team contacts with participants achieved (for ILED and CLED) | 14 week duration of study
Uptake to and continued use of the Oviva® app i.e. percentage of participants willing to try the app and those who continue to use the different app functions over the 12 week period. | 14 week duration of study
Number of other adverse effects potentially associated with the dietary programmes e.g. constipation, fatigue | 14 week duration of study
Number of participants preferring food-based low energy days (for ILED and CLED) | 14 week duration of study
Average time spent by the MDT (for ILED and CLED) | 14 week duration of study
Percentage of contacts with Dietitian conducted face to face after baseline (for ILED and CLED) | 14 week duration of study

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDiarmid S, Harvie M, Aglan A, Winterbottom H, Mubita W, Hulme A, Davies J, Yates J, Krizak S, Perry D, Issa BG. Manchester Intermittent and Daily diet Type 1 Diabetes App Study (MIDDAS-Type 1): protocol for a randomised feasibility trial of an intermittent and continuous low-energy diet in patients with type 1 diabetes and overweight and obesity. BMJ Open. 2023 Jul 20;13(7):e071395. doi: 10.1136/bmjopen-2022-071395. PMID 37474169